CLINICAL TRIAL: NCT03671772
Title: Progression of Prodromal Markers of α-synucleinopathy Neurodegeneration in the First-degree Relatives of Patients With REM Sleep Behavior Disorder: a 5-year Prospective Study
Brief Title: Progression of Prodromal Markers of α-synucleinopathy Neurodegeneration in the FDRs of Patients With RBD
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Zhang Jihui, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 24117018
Record Dates: First submitted 2018-08-30; First posted 2018-09-14 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: REM Sleep Behavior Disorder; Neurodegeneration
Keywords: α-synucleinopathy; Neurodegeneration; Prodromal markers; REM sleep behavior disorder
MeSH Terms: conditions — REM Sleep Behavior Disorder; Nerve Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Thyroid Function Tests(TFT), Vitamin B12, Folate, Complete Blood Count(CBC), Fasting Glucose, Liver Function Tests(LFT), Renal Function Tests(RFT), C-reactive protein(CRP), Fasting lipid, Iron profile, Phosphate, Calcium, Neurosteroid, Genetic analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FDRs of idiopathic RBD patients: First-degree relatives of idiopathic RBD patients
- FDRs of controls: First-degree relatives of controls

SUMMARY:
This study is a prospective study with a mean of 5-year follow-up interval, aims to monitor the progression of α-synucleinopathy neurodegeneration by the evolution of prodromal markers and development of clinical disorders in first-degree relatives (FDRs) of idiopathic REM Sleep Behavior Disorder (RBD) patients and healthy controls.

DETAILED DESCRIPTION:
Idiopathic RBD is implicated as an integral part of progression of α-synucleinopathy neurodegeneration, and patients with idiopathic RBD have increased prevalence of non-motor symptoms (or prodromal markers) closely related to Parkinson's disease(PD). Moreover, the investigator's previous studies have further confirmed the familial aggregation of RBD, and first-degree relatives (FDRs) of RBD patients had more prodromal markers of Parkinson's disease compared with FDRs of healthy controls.

In these regards, current prospective study aims to map the progression and evolution of prodromal markers (including autonomic dysfunction, olfactory loss, color vision impairment, neurocognitive impairment, neuroimaging of dopamine dysfunction, daytime sleepiness and psychiatric disorders), onset of RBD, and neurodegenerative diseases. Finally, other markers, such as physical activity and circadian rhythm and tonic electromyography (EMG) activity level, which have been found to be reliably associated with Parkinson's disease or other neurodegenerative diseases. In this regard, it is also interesting to investigate whether these indicators will additionally predict the progression of prodromal markers of PD.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese aged 40 or above;
2. Being capable of giving informed consent for participation of the study;
3. Sex-matched.

Exclusion Criteria:

1. Younger than 40 years old (as the supposed neurodegenerative process may not have occurred);
2. Not capable of giving informed consent for participation of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants in this proposed study will be recruited from our on-going family cohort of RBD
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Changes of the overall probability of prodromal Parkinson's disease in the FDRs of patients with RBD. | Baseline and 5 years
  Changes of the overall probability of prodromal Parkinson's disease will be calculated based on the Movement Disorder Society (MDS) research criteria for prodromal Parkinson's disease in the FDRs of patients with RBD.

SECONDARY OUTCOMES:
Changes of tonic EMG activity in the FDRs of patients with RBD. | Baseline and 5 years
  Changes of tonic EMG activity is recorded by v-PSG in the FDRs of patients with RBD.
Changes of physical activity level and circadian in the FDRs of patients with RBD. | Baseline and 5 years
  Changes of physical activity level and circadian are recorded by one-week actigraphy in the FDRs of patients with RBD.
New incidence of RBD and α-synucleinopathy in the FDRs of patients with RBD. | Baseline and 5 years
  New incidence of probable RBD, video-polysomnography (v-PSG) confirmed definite RBD and α-synucleinopathies in the FDRs of patients with RBD.

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Zhang, PhD, Principal Investigator — Chinese University of Hong Kong; Yun Kwok Wing, MBChB, Study Director — Chinese University of Hong Kong; Vincent Chung Tong Mok, MBChB, Study Director — Chinese University of Hong Kong; Shirley Xin Li, PhD, Study Director — Hong Kong University
Locations (1):
- Department of psychiatry, Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Researcher in other sleep centers are also conducting similar study, there may be a plan for further collaboration on sharing the database